CLINICAL TRIAL: NCT02961998
Title: Preventive Effect of Celecoxib on Sorafenib-related Hand Foot Syndrome
Brief Title: Preventive Effect of Celecoxib on Sorafenib-related Hand Foot Syndrome, a Single Center, Randomized Controlled Clinical Trail
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongguo Zhou, Associate Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-FXY-006
Record Dates: First submitted 2016-11-06; First posted 2016-11-11 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; sorafenib; celecoxib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Celecoxib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Celecoxib group (Experimental): Patients were treated with sorafenib taking capsules celecoxib (Celebrex) at the same time, 200mg/day, last 6 months
  Interventions: Drug: Celecoxib; Drug: Sorafenib
- Control group (Active Comparator): Patients take sorafenib only.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Celecoxib — Patients from experimental group will take celecoxib, except for sorafenib
  Arms: Celecoxib group
Drug: Sorafenib — Each group will receive sorafenib as basic treatment.

SUMMARY:
Hepatocellular carcinoma (HCC) is a common fatal malignant tumor, although with the popularity of health examination, most patients were diagnosed as HCC in advanced stages so far. Sorafenib is currently recognized worldwide as the only effective treatment for advanced HCC. However, sorafenib need long-term medication, and will bring a series of side effects, including, hand, foot and comprehensive syndrome (Hand-foot syndrome, HFS) limbs swelling, rash, peeling, pain.Occurrence rate of HFS is about 21%-51%, which seriously affect patient's quality of life.Besides, this side effects appeared to be dose-related.When severe HFS happened, sorafenib need to reduce dosage or discontinue administration, which could seriously affect the patient's survival. Therefore, investigators designed this prospective randomized controlled study to explore preventive effect of celecoxib for sorafenib related HFS, the influence on the quality of life in patients with, and also the synergistic anti-tumor effect of celecoxib in combination with sorafenib on HCC. This study will explore horizon of improving treatment for sorafenib in patients with advanced HCC,quality of life and tumor control.

ELIGIBILITY:
Inclusion Criteria:

* 1.Diagnosed with HCC according to the Primary liver cancer diagnosis and treatment practices published by the Ministry of Health in 2011 China
* 2.A Karnofsky Performance Status (KPS) score ≥70 points
* 3.Age between 18 and 70 years
* 4.Child-Pugh classA or B (class B patients had scores no greater than 7 points). In addition, the baseline laboratory tests had to meet the following criteria: white blood cells (WBCs) ≥1.5 × 109/L, platelets ≥50 × 109/L, hemoglobin ≥80 g/L, serum aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2 x the upper limit of normal (ULN), serum creatinine ≤ 1.5 x ULN, an international normalized ratio (INR)<1.5 or prothrombin time < the ULN + 4 seconds, albumin ≥30 g/L, and total bilirubin ≤34mmol/L
* 5.Patients with advanced hepatocellular carcinoma who failed first-line therapy with surgery，radiofrequency ablation

Exclusion Criteria:

* 1.Pugh Child-Pugh Grade C, or with massive ascites or had a history of hepatic encephalopathy, or previous history of gastrointestinal bleeding
* 2.Poor general condition or cachexia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incidence of participants with clinically definite Sorafenib-related Hand Foot Syndrome | within the first 6 months after sorafenib administration

SECONDARY OUTCOMES:
Overall survival | one year

CONTACTS AND LOCATIONS:
Overall Officials: Minshan Chen, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen JC, Wang JC, Pan YX, Yi MJ, Chen JB, Wang XH, Fu YZ, Zhang YJ, Xu L, Chen MS, Zhang RX, Zhou ZG. Preventive effect of celecoxib in sorafenib-related hand-foot syndrome in hepatocellular carcinoma patients, a single-center, open-label, randomized, controlled clinical phase III trial. Am J Cancer Res. 2020 May 1;10(5):1467-1476. eCollection 2020. PMID 32509392